CLINICAL TRIAL: NCT03450694
Title: Role of Ultrasound in Diagnosis of Laryngeal Lesions
Brief Title: Role of Ultrasound in Laryngeal Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennat-Alllah Samy Abdelaziz, mennat-Allah Samy, Assiut University
Other Study IDs: US in laryngeal lesions
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Laryngeal Disease
MeSH Terms: conditions — Laryngeal Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound — ultrasound is a non-invasive and not expensive method, availiable at almost all institutions.

SUMMARY:
The aim of the study is to assess the efficiency and limitations of ultrasound in detecting and characterizing laryngeal anatomy and study of some laryngeal disorders and their ultrasonographic appearance.

DETAILED DESCRIPTION:
The larynx contains the vocal cords and serves as the opening to the tracheobronchial tree. Laryngeal lesions include: benign laryngeal tumors, contact ulcers, laryngitis, laryngeoceles, malignant laryngeal tumors, spasmodic dysphonia, vocal cord paralysis, vocal cord polyps, nodules and granulomas.

Laryngeal cancers account for about one quarter of all head and neck cancers, most of which affect the true vocal cords. Black men are affected more commonly than white men. The male to female incidence ratio is about 4:1.

Laryngeal cancer is the 19th most common cause of cancer death worldwide, with around 83,400 deaths from laryngeal cancer in 2012 (1% of total cancer deaths). Cancer of larynx is one of the most common malignancies in Europe, with about 52,000 new cases per year. The yearly incidence rate in Europe is about 8 per 100,000.

Different methods were used successfully for the diagnosis of many laryngeal diseases. Rigid endoscope was used for laryngeal evaluation with the advantage that the image is large, bright and clear which allows early diagnosis of the lesion (Shao et al, 2002).

Unfortunately, not all patients can tolerate the laryngoscope especially those with a sensitive gag reflex, patients with limit of jaw or neck mobility or patients suffering from stridor. It is also difficult in most infants and children .

Even during laryngoscopy the exact extension of laryngeal tumor, its infiltration and invasion of the laryngeal skeleton can sometimes be hard to assess. Thus, laryngoscopy alone may not be sufficient in some cases to judge the extent of infiltrative processes or measure the exact infiltration of a tumor. For this reason computed tomography (C.T) as well as magnetic resonance imaging (MRI) is often used to supplement laryngoscope as an additional imaging tool in the estimation of tumor extension and size.

Ultrasonography is a non-invasive modality, available at almost all institutions, not expensive, easily reproducible method of examining the larynx in infants and children, can be used safely during pregnancy in contrast to scan, portable and can be easily transferred to patients with difficult mobilization.

Ultrasound became a very important, widely used diagnostic tool for head and neck diseases; however, it was rarely used in the diagnosis of laryngeal diseases. This was because of the problem in visualization of laryngeal structures and thus in performing a complete laryngeal sonographic examination due to the acoustic extinction of the ultrasound by the ossified laryngeal cartilages .

Researchers have recently used color Doppler imaging to study the surface mucosal waves of the vocal folds. During the last several years high-frequency ultrasound became an effective diagnostic tool with small, flexible ultrasound transducers .

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of laryngeal lesions in adult age group between age 18:65 years of both sexes.

Exclusion Criteria:

* patients < 18 years
* patients > 65 years
* patients with spinal lesions who needs spinal immobilization

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients complaining of laryngeal lesions in adult adult age group between 18:65 years of both sexes. they are previously diagnosed by laryngoscope.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
role of ultrasound in diagnosis of laryngeal lesions | baseline
  statistical study will be done between ultrasound and laryngoscope to assess sensitivity, specificity and accuracy of ultrasound in detecting lesions, differentiate benign from malignant lesions and reach final diagnosis of the laryngeal lesions.

REFERENCES:
- [Background] Agrawal N, Ha PK. Management of early-stage laryngeal cancer. Otolaryngol Clin North Am. 2008 Aug;41(4):757-69, vi-vii. doi: 10.1016/j.otc.2008.01.014. PMID 18570957
- [Background] 3. Arruti, A. and Poumayrac, D.M., 2010. Larynx ultrasonography: an alternative technique in the evaluation of the aero-digestive crossroad. Rev Imagenol, 14(1), pp.30-6.
- [Background] American Cancer Society, 2008. Cancer facts & figures. The Society.
- [Background] Arens C, Eistert B, Glanz H, Waas W. Endolaryngeal high-frequency ultrasound. Eur Arch Otorhinolaryngol. 1998;255(5):250-5. doi: 10.1007/s004050050052. PMID 9638467
- [Background] Muscat JE, Liu HP, Livelsberger C, Richie JP Jr, Stellman SD. The nicotine dependence phenotype, time to first cigarette, and larynx cancer risk. Cancer Causes Control. 2012 Mar;23(3):497-503. doi: 10.1007/s10552-012-9909-x. Epub 2012 Feb 25. PMID 22367700
- [Background] Shao J, Stern J, Wang ZM, Hanson D, Jiang J. Clinical evaluation of 70 degrees and 90 degrees laryngeal telescopes. Arch Otolaryngol Head Neck Surg. 2002 Aug;128(8):941-4. doi: 10.1001/archotol.128.8.941. PMID 12162775
- [Background] Shau YW, Wang CL, Hsieh FJ, Hsiao TY. Noninvasive assessment of vocal fold mucosal wave velocity using color doppler imaging. Ultrasound Med Biol. 2001 Nov;27(11):1451-60. doi: 10.1016/s0301-5629(01)00453-7. PMID 11750743
- [Background] Torre LA, Siegel RL, Ward EM, Jemal A. Global Cancer Incidence and Mortality Rates and Trends--An Update. Cancer Epidemiol Biomarkers Prev. 2016 Jan;25(1):16-27. doi: 10.1158/1055-9965.EPI-15-0578. Epub 2015 Dec 14. PMID 26667886
- [Background] 12. Wendy, D., 2007. Laryngeal ultrasound provides non invasive assessment of vocal fold lesions. Ann Otol Rhinol Laryngol, 171, pp.631-647.
- [Background] Wolf M, Primov-Fever A, Amir O, Jedwab D. The feasibility of rigid stroboscopy in children. Int J Pediatr Otorhinolaryngol. 2005 Aug;69(8):1077-9. doi: 10.1016/j.ijporl.2005.03.004. Epub 2005 Mar 31. PMID 16005350